CLINICAL TRIAL: NCT07234136
Title: Cholecystectomy TIming for Mild Acute Biliary Pancreatitis [CTIMAP]: a Società Lombarda di Chirurgia Observational Study
Acronym: CTIMAP
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marcello Maestri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: CTIMAP
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Mild Acute Biliary Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Mild Acute Biliary Pancreatitis treated with the Same Admission Cholecystectomy
- Patients with Mild Acute Biliary Pancreatitis treated with Interval Cholecystectomy

SUMMARY:
CTIMAP is a prospective multicenter observational study on patients with Mild Acute Biliary Pancreatitis (MABP) treated with Same Admission Cholecystectomy (SAC) and Interval Cholecystectomy (IC). The rationale of this study is to investigate the timing of cholecystectomy after MABP applied by Lombard surgeons and compare SAC and IC, with the hypothesis that SAC would reduce the risk of recurrent Gallstones Related Events (GRE) without increasing the difficulty of surgery and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* to be admitted with a diagnosis of acute pancreatitis, as defined according to 2012 Atlanta Criteria
* pancreatitis is mild as defined according to 2012 Atlanta Criteria
* the etiology of pancreatitis is a gallstone related (finding of stones or sludge in the gallbladder on in the main biliary duct)
* be greater than or equal to 18 years old
* provide signed and dated informed consent form
* willing to comply with all study procedures and be available during the study

Exclusion Criteria:

* pregnancy or lactation
* pancreatitis not related to a gallstone etiology
* chronic pancreatitis
* moderately severe or severe pancreatitis
* alcohol abuse
* anything that would place the individual at increased risk or prevent the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MABP treated with SAC or IC
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of 6-month readmission due to GRE after hospitalization for MABP | 6 months

SECONDARY OUTCOMES:
30-day postoperative complications rate after SAC and after IC in patients with MABP | Day 30
30-day postoperative biliary complications rate after SAC and after IC in patients with MABP | Day 30
30-day postoperative mortality rate after SAC and after IC in patients with MABP | Day 30
Intraoperative complication rate during SAC and IC | Day of SAC or IC
Rate of bail out procedures during SAC and IC | Day of SAC or IC
Conversion to open laparotomy rate during SAC and during IC in patients with MABP | Day of SAC or IC
Operative times (minutes) of SAC and of IC in patients with MABP | Day of SAC or IC
Postoperative length of stay (PO-LOS) after SAC and after IC in patients with MABP | At discharge
Total length of stay (T-LOS) of patients with MABP treated with SAC and with IC | At discharge
Rate of patients who after six months after discharge did not receive cholecystectomy (no-cholecystectomy group) | 6 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy